CLINICAL TRIAL: NCT05752773
Title: Risk Identification and Prediction of Myocardial Injury After Laparoscopic Pheochromocytoma/Paraganglioma Resection:A Ambispective Cohort Study.
Brief Title: Prediction of Myocardial Injury After Laparoscopic Pheochromocytoma/ParaGangLioma Resection
Acronym: MI-PPGL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lan Ling, Attending doctor, Peking Union Medical College Hospital
Other Study IDs: 2022-PUMCH-B-0071
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: PGL
Keywords: myocardial injury; prediciton; pheochromocytoma/paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study was conducted in patients undergoing elective laparoscopic pheochromocytoma/paraganglioma(PPGL) resection. It mainly answers the following two main questions:

1. What are the risk factors for myocardial injury after laparoscopic PPGL resection？
2. How to establish the myocardial injury prediction model of laparoscopic PPGL resection?

Participants were not required to perform additional research work other than the usual postoperative follow-up within 30 days after surgery. No control group was set in this study, and no additional clinical intervention was performed.

DETAILED DESCRIPTION:
MI-PPGL is a single-center observational ambispective cohort study.On the basis of retrospective study, the research team plans to build a structured database to investigate the incidence of myocardial injury in laparoscopic PPGL-resection, and further analyze myocardial injury related risk factors. In particular, timing data such as vital signs(blood pressure,heart rate)will be included to construct an efficient and robust myocardial injury prediction model. At the same time, a prospective cohort study is carried out to verify the model, so as to test the prediction ability of myocardial injury and reduce the incidence of myocardial injury.

The investigators expect to enroll 700 patients, including at least 550 patients retrospectively and 150 patients prospectively.In this study, the main endpoint events of the prediction model are binary outcome. Conservatively estimated according to the "10EPV" principle, that is, each predictive factor included in the model needs at least 10 positive outcome endpoint for estimation (10 events per variable). The investigators expected 5 to 8 predictors to be included in the model, and at least 80 positive events to be included. The incidence of perioperative myocardial injury is 12~20%, so the estimated sample size was at least 666 patients. Considering the absence of data or subject withdrawal from the study. so the investigators expected to include 700 patients, including at least 550 retrospectively and 150 prospectively.

STATA (version 15.0; Stata Corp., TX, USA) and R 3.6.1 software (R Foundation for Statistical Computing, Vienna, Austria) will be used for statistical analysis. Binary logistic regression was used to screen risk factors and stratify risk levels. P<0.05 was considered statistically significant. For predictive modeling, clinical databases were 9:1 or 8: 2. Randomly split into training samples and verification samples. In the training samples, optimal subset method and LASSO regression will be used for feature selection.Receiver operating characteristic curve (ROC curve) was used to represent the model differentiation, and Nomogram was used to represent the predictive factors of multiple logistic regression. In the verification samples, Hosmer-Lemeshow goodness of fit test was used to test the calibration degree of the model, and P>0.05 was the acceptable level of estimated fitting of the model. Decision curve analysis (DCA curve) was used to verify the clinical applicability.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for Laparoscopic PPGL resection

Exclusion Criteria:

1. Open or laparoscopic conversion to open PPGL resection was excluded
2. Cardiac paraganglioma was excluded
3. History of congenital heart disease or cardiac surgery was excluded
4. Patients with preoperative troponin/hypersensitive troponin elevation were excluded
5. Carotid body tumor and accessory ganglioma of jugular tympanum without endocrine function were excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2013 to May 2025, adult patients underwent elective laparoscopic PPGL resection.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial injury after laparoscopic PPGL resection | 30days after surgery
  Myocardial injury was defined as an elevated troponin I level exceeding the 99th percentile upper reference limit due to cardiac ischemic causes.

SECONDARY OUTCOMES:
Acute myocardial infarction | 30days after surgery
  An increase in troponin exceeding 99% of the reference limit is associated with at least one of the following: 1. Symptoms of myocardial ischemia; 2. New ECG ischemic changes (ST elevation or depression or abnormal Q wave; 3. Imaging findings of abnormal new ventricular wall movement or loss of viable myocardia consistent with ischemic etiology; 4. Coronary thrombosis was confirmed by coronary intervention (angiography) or autopsy.
Nonfatal cardiac arrest | 30days after surgery
  An event in which cardiac activity abruptly stops, usually through CPR and/or defibrillation or cardioversion, or cardiac pacing reversal, resulting in a loss of normal signs of breathing and spontaneous circulation.
Congestive heart failure | 30days after surgery
  Patients with new postoperative symptoms and signs: fatigue, dyspnea, upright breathing, paroxysmal dyspnea at night, increased jugular vein pressure, wet rales found on physical examination, heart enlargement, pulmonary vascular congestion.
New atrial fibrillation | 30days after surgery
  new atrial fibrillation heart rate confirmed by electrocardiogram or color Doppler ultrasound after surgery.
Stroke | 30days after surgery
  CT or MRI showing cerebral infarction or cerebral hemorrhage or new neurological symptoms (hemiplegia, decreased muscle strength, or dysphonia) lasting more than 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: LING LAN, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital,Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lan L, Ma Y, Zhao Y, Li Y, Zhang Y, Shen L, Zhang Y, Huang Y. Prediction of postoperative myocardial injury in patients undergoing laparoscopic pheochromocytoma/paraganglioma resection: protocol for an ambispective cohort study. BMJ Open. 2025 Feb 7;15(2):e091975. doi: 10.1136/bmjopen-2024-091975. PMID 39920072